CLINICAL TRIAL: NCT03877549
Title: Dexamethasone Administered Via the Epidural Catheter as an Adjunct in Patients Undergoing Cesarean Delivery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left Henry Ford Health before completion.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Katherine Nowak, Research Manager, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12391
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain
Keywords: dexamethasone; labor epidural; cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): 10cc 0.0625% bupivacaine
  Interventions: Drug: Dexamethasone
- Low Dose (Experimental): 4mg Dexamethasone + 10cc 0.0625% bupivacaine
  Interventions: Drug: Dexamethasone
- Higher Dose (Experimental): 8mg Dexamethasone + 10cc 0.0625% bupivacaine
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Additional of two different doses of dexamethasone via the epidural catheter during surgical closure after cesarean section

SUMMARY:
This study will evaluate the ability of dexamethasone to enhance labor epidurals when administered as an adjunct to local anesthetics via an epidural catheter. Patients undergoing elective cesarean sections will be randomized into three groups, each receiving the same combined spinal epidural (CSE). At surgical closure, Group 1 will receive 10cc bupivacaine 0.0625%, Group 2 will receive 10cc bupivacaine 0.0625% +4mg dexamethasone, and Group 3 will receive 10cc bupivacaine 0.0625% + 8mg dexamethasone (4mg). VAS, sedation, nausea, and satisfaction scoring will be measured on patient follow-up to compare the outcomes of the different treatment groups.

DETAILED DESCRIPTION:
This study will evaluate the ability of dexamethasone to enhance labor epidurals when administered as an adjunct to local anesthetics via an epidural catheter. Patients undergoing elective cesarean sections will be randomized into three groups using a random allocation table. Group assignment will be performed by opening a previously prepared numbered opaque envelope containing the assignment. Each group will receive the same combined spinal epidural (CSE) containing 10-12mg hyperbaric bupivacaine, 150mcg preservative-free morphine, and 15mcg fentanyl. At surgical closure, Group 1 will receive 10cc bupivacaine 0.0625%, Group 2 will receive 10cc bupivacaine 0.0625% +4mg dexamethasone, and Group 3 will receive 10cc bupivacaine 0.0625% + 8mg dexamethasone (4mg). In order to maintain this as a double-blinded study, the patient will not be told which medication was administered and the drug will be given by one anesthesiologist and the patient follow-up will be performed by a different anesthesiologist. VAS, sedation, nausea, and satisfaction scoring will be measured on patient follow-up to compare how these outcomes compare between the different treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Parturients in their 3rd trimester who are receiving a planned cesarean delivery
* Primiparous and multiparous pregnancies
* American Society of Anesthesia (ASA) classes 1, 2 , and 3

Exclusion Criteria:

* Patients for whom neuraxial anesthesia was either declined, unsuccessful, or contraindicated
* Gestational Diabetics
* Diabetics
* Patients allergic to dexamethasone, local anesthetics, or opioids
* Patients that are immunosuppressed
* Patient who received systemic steroids within the preceding 48 hours

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Scores | up to 48 hours post-op
  Visual Analog Scale for Pain, uses the Wong-Baker method of presenting faces with different reactions to pain and scales the patient based on the patient selection of a face. The range goes from 0-10. 0 is pain-free and 10 is excruciating pain.

SECONDARY OUTCOMES:
Nausea/ Vomiting Scale | up to 48 hours post-op
  Baxter Retching Faces. (BARF) pictorial faces of someone wrenching that is used to scale a patient nausea and vomiting. The range goes from 0-10. 0 is nausea-free and 10 is intractable nausea and vomiting.
Pruritus Score | up to 48 hours post-op
  Pruritus Scale is also a visual analog scale that has a patient rate their discomfort on a number line that gradates the severity.
Sedation Score | up to 48 hours post-op
  Richmond Agitation and Sedation Scale (RASS). Its a well known and utilized scale that gradates a patients level of sedation based on various responses to stimuli. The Score goes from -4 to +5. -4 represents a combative and violent patient and +5 represents a patient unresponsive to physical stimuli.
Motor Function | up to 48 hours post-op
  Bromage scale is a scoring system that assesses lower extremity motor function based on ones ability to flex and extend various parts of the leg. Score is 1-4. 1 is no motor block and 4 is complete motor block.
Satisfaction Score | up to 48 hours post-op
  Customer Satisfaction score (CSAT) is a scoring system that scores satisfaction on a 1-5 basis. 1 is very unsatisfied and 5 is very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States